CLINICAL TRIAL: NCT00420680
Title: A Multi -Center, Randomized, Parallel-Group, Placebo-Controlled, Safety Assessor-Blinded Trial, Evaluating the Safety and Efficacy of Sugammadex in Cardiac Patients
Brief Title: Safety and Efficacy Evaluation of Sugammadex in Cardiac Patients (19.4.309)(P05934)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05934; EudraCT Number: 2005-002000-42; 19.4.309
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Sugammadex 2.0 mg/kg
  Interventions: Drug: Sugammadex
- Arm 2 (Experimental): Sugammadex 4.0 mg/kg
  Interventions: Drug: Sugammadex
- Arm 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sugammadex — Sugammadex, 2.0 mg/kg given as a reversal agent at reappearance of T2 after 0.6 mg/kg rocuronium
  Other Names: Org 25969
  Arms: Arm 1
Drug: Sugammadex — Sugammadex, 4.0 mg/kg given as a reversal agent at reappearance of T2 after 0.6 mg/kg rocuronium.
  Other Names: Org 25969
  Arms: Arm 2
Drug: Placebo — Placebo given at reappearance of T2 after 0.6 mg/kg rocuronium
  Arms: Arm 3

SUMMARY:
The purpose of this study is to evaluate the safety of 2.0 mg/kg and 4.0 mg/kg sugammadex given as a reversal agent at reappearance of T2 after 0.6 mg/kg rocuronium in cardiac patients

ELIGIBILITY:
Inclusion Criteria:

* Cardiac patients of NYHA Class II to III
* ASA class maximally 4
* Age at least 18
* Scheduled for elective, non-cardiac surgery under general anesthesia with propofol in the supine position, with planned muscle relaxation using rocuronium and allowing for 12-lead ECG assessment during surgery;
* Given written informed consent.

Exclusion Criteria:

* Disorders interfering with the reliability of the assessments (e.g. ECG measurements), such as paroxysmal atrial fibrillation or the presence of a pacemaker
* Known or suspected neuromuscular disorders impairing NMB
* Known or suspected significant renal dysfunction
* Known or suspected (family) history of malignant hyperthermia
* Known or suspected allergy to narcotics, muscle relaxants or other medication used during general anesthesia
* Intended) use of medication expected to interfere with the effect of rocuronium as given in this trial, based on the dose and/or the time of administration (such as antibiotics, anticonvulsants and Mg2+ )
* Pregnancy (pregnancy to be excluded for women both from medical history and by an hCG test within 24 h before surgery, except for women who were not of childbearing potential, i.e. at least 2 years menopausal or have undergone tubal ligation or a hysterectomy)
* Childbearing potential without using any method of birth control or using only hormonal contraception as birth control (subjects were allowed to participate if they were willing to use a condom, or a diaphragm with spermicide, or IUD, or have a vasectomized partner (>6 months) or abstinence, for one month after participation in the trial)
* Breast -feeding
* Prior participation in any trial with Org 25969
* Participation in another clinical trial not pre -approved by Organon, within 30 days of entering into trial 19.4.309

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-11-07 (Actual); Primary Completion 2006-08-01 (Actual); Study Completion 2006-08-01 (Actual)

PRIMARY OUTCOMES:
to evaluate the safety of 2.0 and 4.0 mg/kg sugammadex in cardiac patients compared to placebo | after surgery

SECONDARY OUTCOMES:
to evaluate the time to recovery from a neuromuscular block induced by rocuronium after reversal at reappearance of T2 by 2.0 and 4.0 mg/kg sugammadex in cardiac patients | after surgery

REFERENCES:
- [Result] Dahl V, Pendeville PE, Hollmann MW, Heier T, Abels EA, Blobner M. Safety and efficacy of sugammadex for the reversal of rocuronium-induced neuromuscular blockade in cardiac patients undergoing noncardiac surgery. Eur J Anaesthesiol. 2009 Oct;26(10):874-84. doi: 10.1097/EJA.0b013e32832c605b. PMID 19455040
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html